CLINICAL TRIAL: NCT00523783
Title: 24-Week Naturalistic Observational Study of Efficacy of Quetiapine in Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Seroquel Long-Term NIS for Schizophrenia Patients
Acronym: SELECT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-NKR-SER-2007/1
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2007-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective; quetiapine; long-term efficacy; Naturalistic; Observational
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the efficacy of 24-week treatment with quetiapine in patients with schizophrenia or schizoaffective disorder

ELIGIBILITY:
Inclusion Criteria:

* The patient and the patient's legal representative (if any) must understand the nature of the study and must have given written consent
* The patient suffers from schizophrenia or schizoaffective disorder according to DSM-IV-TR
* The patient is between 18 and 65 years old(extremes included)
* On the basis of physical and neurological examination, medical history, the patient is, in the investigator's opinion, otherwise healthy
* If the subject is a female of childbearing potential, she must be not pregnant or breast-feeding and be using a reliable method of contraception. Reliable methods may include abstinence, hormonal contraceptives (eg,oral contraceptives or long-term injectable or implantable hormonal contraceptives), double-barrier methods (eg, condom and diaphragm, condom and foam, condom and sponge), intrauterine devices, and tubal ligation

Exclusion Criteria:

* The patients who have known hypersensitivity to quetiapine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-11 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Woo Bahn, Study Director — AstraZeneca Korea
Locations (3):
- South Korea (3):
  - Research Site, Seoul, Dongdamoon-gu
  - Research Site, Seoul, Kangnam-gu
  - Research Site, Seoul, Songpa-gu